CLINICAL TRIAL: NCT05261451
Title: Effectiveness of Occupational Therapy Trauma Informed Workshops and Consultations for Teachers at Head Start
Brief Title: Occupational Therapy Trauma Informed Workshops and Consultations for Teachers at Head Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Arezou Salamat, Principal Investigator, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5210415
Record Dates: First submitted 2022-02-14; First posted 2022-03-02 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Trauma
Keywords: occupational therapy; trauma informed care
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Head Start Teachers (Experimental): Participants will engage in three 1- hour workshops and optional consultations with an occupational therapist
  Interventions: Other: Workshop

INTERVENTIONS:
Other: Workshop — Participants will engage in three 1 hour workshops about trauma informed care. They will complete pre and post measure before engaging in the workshops

SUMMARY:
This study will utilize a pre/post mix method design

Quantitative data will be gathered through surveys (including satisfaction questionnaires) administered pre/post workshops.

Qualitative data will be obtained through interviews post- workshop and consultations.

ELIGIBILITY:
Inclusion Criteria:

* Home Visitors or Teaching Staff at Head Start within San Bernardino County
* Between 18-65 years of age
* All genders
* English Speaking

Exclusion Criteria:

* NA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Post-Survey | Within 1 week after the consultations
  knowledge and experience
  knowledge and experiences gained related to early childhood trauma. Higher scores indicate greater knowledge

SECONDARY OUTCOMES:
Interview | Within 2 weeks after the consultations
  Post interviews will be completed with participants who also complete the consultations

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No